CLINICAL TRIAL: NCT01930799
Title: Bladder Management in Patients With Multiple Sclerosis: Optimizing Practice Patterns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GMA-NDO-112
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Sclerosis; Urinary Bladder Diseases
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Enrolled Patients (Other): Site will implement a systematic approach to screening bladder health dysfunction in multiple sclerosis patients, providing bladder health management education, and initiating appropriate urologist referrals.
  Interventions: Behavioral: Systematic Screening and Education Regimen

INTERVENTIONS:
Behavioral: Systematic Screening and Education Regimen — Site will implement a systematic approach to screening bladder health dysfunction in multiple sclerosis patients, providing bladder health management education, and initiating appropriate urologist referrals.

SUMMARY:
This study will assess the impact of a systematic bladder health screening and disease education regimen as well as the implementation of a referral process on the quality of life of multiple sclerosis patients with bladder dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting multiple sclerosis and currently being treated by study doctor

Exclusion Criteria:

* Diagnosis of primary-progressive, secondary-progressive, or progressive-relapsing multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Fresno, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Enrolled Patients
Started | 120
Completed | 112
Not Completed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Patients
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the King's Health Questionnaire (KHQ) Domain Scores
Description: The KHQ is a valid and reliable patient reported outcome measure for the assessment of quality of life in subjects with urinary incontinence that contains the following 8 domains: general health perception, incontinence impact, role limitations, physical limitations, social limitations, personal relations, emotions, sleep/energy, and severity measures. The KHQ domain scores are based on a scale of 0-100, with a lower score indicating less severity. Decreases in KHQ domain scores indicate an improvement in quality of life and increases in KHQ domain scores indicate a worsening in quality of life.
Time Frame: Baseline, Month 6
Population: Eligible and enrolled subjects who completed the Month 6 visit
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | All Enrolled Patients
Number analyzed (Participants) | 112
Scores on a Scale
  Baseline (BL)-General Health Perception | 39.7 (23.1)
  Chng from BL at M6-General Health Percept (N=111) | 2.5 (22.3)
  BL-Incontinence Impact | 60.7 (23.8)
  Chng from BL at M6-Incontinence Impact (N=111) | 1.2 (24.2)
  BL-Role Limitations (N=111) | 43.8 (29.6)
  Chng from BL at M6-Role Limitations (N=111) | -6.9 (27.5)
  BL-Physical Limitations (N=111) | 45.3 (28.0)
  Chng from BL at M6-Physical Limitations (N=111) | -9.8 (26.3)
  BL-Social Limitations (N=110) | 31.7 (28.6)
  Chng from BL at M6-Social Limitations (N=110) | -9.0 (24.5)
  BL-Personal Relations (N=85) | 25.9 (30.3)
  Chng from BL at M6-Personal Relations (N=78) | -9.0 (24.9)
  BL-Emotions | 35.7 (28.4)
  Chng from BL at M6-Emotions | -9.0 (21.8)
  BL-Sleep/Energy | 41.7 (27.8)
  Chng from BL at M6-Sleep/Energy | -8.2 (25.1)
  BL-Severity Measures | 46.9 (23.7)
  Chng from BL at M6-Severity Measures | -5.7 (17.7)

2. Secondary Outcome: Percentage of Patients Who Agree/Completely Agree With Each Question on the Patient Post-Video Questionnaire
Description: The Patient Post-Video Questionnaire was based on 5 individual questions assessing the patient's perception of the utility of the video in helping them 1) understand how MS can affect the bladder, 2) how to recognize bladder symptoms, 3) understand various treatment options, 4) understand self-help strategies, and 5) better manage their bladder problems. Percentages represent the proportion of patients who "agree/completely agree" with each question. Patients viewed the video at the Baseline visit, then completed the Patient Post-Video Questionnaire immediately after viewing the video at the Baseline visit.
Time Frame: Baseline
Population: Eligible enrolled subjects
Measure: Number; unit: Percentage of Patients
Arm/Group | All Enrolled Patients
Number analyzed (Participants) | 117
Percentage of Patients
  Understand how MS can affect the bladder | 94.0
  How to recognize bladder symptoms | 94.0
  Understand various treatment options | 94.0
  Understand self-help strategies | 88.9
  Better manage their bladder problems | 81.2

ADVERSE EVENTS:
Description: Adverse events and serious adverse events were not collected, as no treatment was administered in this study. This study evaluated the use of an educational video.
Arm/Group | All Enrolled Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.